CLINICAL TRIAL: NCT02628613
Title: Phase II Randomized Clinical Trial and Biomarker Analysis of Paclitaxel Plus Epirubicin Versus Vinorelbine Plus Epirubicin as Neoadjuvant Chemotherapy in Locally Advanced HER2-Negative Breast Cancer With TEKT4 Variations
Brief Title: Neoadjuvant Paclitaxel Plus Epirubicin Versus Vinorelbine Plus Epirubicin in Breast Cancer With TEKT4 Variations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, MD, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20150309
Record Dates: First submitted 2015-12-05; First posted 2015-12-11 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Neoadjuvant chemotherapy; TEKT4
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Epirubicin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel plus Epirubicin (Active Comparator): Paclitaxel plus Epirubicin for 4 cycles, paclitaxel 80 mg/m2 IV on day 1, 8 and 15, epirubicin 90 mg/m2 IV on day 1, and dosing interval is 21 days.
  Interventions: Drug: Paclitaxel plus Epirubicin
- Vinorelbine plus Epirubicin (Experimental): Vinorelbine plus Epirubicin for 4 cycles, vinorelbine 25 mg/m2 IV on day 1, 8 and 15, epirubicin 90 mg/m2 IV on day 1, and dosing interval is 21 days.
  Interventions: Drug: Vinorelbine plus Epirubicin

INTERVENTIONS:
Drug: Vinorelbine plus Epirubicin — Evaluate the efficiency and safety of vinorelbine plus epirubicin as neoadjuvant chemotherapy in locally advanced HER2-negative breast cancer with TEKT4 variations
  Arms: Vinorelbine plus Epirubicin
Drug: Paclitaxel plus Epirubicin — standard neoadjuvant chemotherapy
  Arms: Paclitaxel plus Epirubicin

SUMMARY:
The purpose of this study is to compare the efficiency and safety between paclitaxel combined with epirubicin and vinorelbine combined with epirubicin when used in neoadjuvant chemotherapy for locally advanced (IIb-IIIc) HER2-negative breast cancer with TEKT4 variations.

DETAILED DESCRIPTION:
Taxane-based chemotherapy is the cornerstone treating breast cancer, however remarkable percentage of breast cancer patients presents with primary or secondary taxane resistance. Currently no established biomarker has been reported clinically for predicting taxane sensitivity. Our previous study indicated that TEKT4 variation decreased the stability of intracellular microtubule, and TEKT4 variant cells behaves higher resistance to microtubule-stabilizing agents such as taxane, while enhanced sensibility to microtubule depolymerization agents such as vinorelbine. This study is intended to confirm that TEKT4 variation predicts the prognosis of taxane-based chemotherapy through the prospective clinical trials.

This study intends to evaluate the efficiency and safety of two neoadjuvant therapies: paclitaxel combined with epirubicin and vinorelbine combined with epirubicin, in treating locally advanced (IIb-IIIc) HER2-negative breast cancer with TEKT4 variation.

Primary endpoint of study: pathologic Complete Response (pCR). Secondary endpoints of the study: Objective response rate (CR+PR). Exploratory endpoint: Based on pretreatment tumor and matched blood samples, the correlation between biomarker and efficiency is explored.

This open single center prospective randomized control study includes patients locally advanced (IIb-IIIc) HER2-negative patients with TEKT4 variation diagnosed with histopathology and Sanger sequencing. Patients randomized to Group A or Group B to receive respective neoadjuvant chemotherapy. Among which Group A: PE x 4 cycles (paclitaxel + epirubicin), paclitaxel: 80 mg/m2 IV on day 1, 8 and 15; epirubicin: 90 mg/m2 IV on day 1, and dosing interval is 21 days. Group B: NE x 4 cycles (vinorelbine + epirubicin), vinorelbine: 25 mg/m2 IV on day 1, 8 and 15; epirubicin: 90 mg/m2 IV on day 1, and dosing interval is 21 days.

Patients of both groups were performed with diagnostic puncture before treatment and over half of treatment course in order to obtain information about dynamic change of Ki67 and other parameters; Surgery will be performed after 4 cycles of chemotherapy, followed with subsequent adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years old
2. Expected survival > 12 months
3. Baseline ECOG Performance Status rating 0-1
4. Naïve to chemotherapy or hormonal treatments
5. Radiologically confirmed and biopsy diagnosed invasive ductal carcinoma of breast and prepared to be treated surgically
6. Locally advance breast cancer of stage IIb-IIIc
7. HER-2 negative confirmed by immunohistochemistry, Ki-67≥20%
8. TEKT4 variation confirmed by DNA sequencing
9. No concurrent malignancy (except controlled cervical carcinoma in situ or basal cell carcinoma of skin)
10. Patients have measurable lesions (according to RECIST v1.1 criteria)
11. Intention to cooperate with baseline puncture and neoadjuvant therapy
12. No advanced metastasis or metastasis involving brain or liver
13. Adequate bone marrow function, blood routine examination shows neutrophil count ≥ 1.5x109/L, hemoglobin level ≥ 100 g/L, Platelets ≥ 100 x 109/L
14. Adequate liver and kidney function, serum aminotransferase (AST) ≤ 60U/L, serum total bilirubin ≤ 2.5 times ULN, serum creatinine ≤110μmol/L, urea nitrogen ≤7.1mmol/L
15. No coagulation abnormality
16. Normal heart function, with normal ECG and LVEF ≥ 55%
17. Women of childbearing age agree to take reliable contraceptive measures during clinical trials, and negative serum or urine pregnancy test within 7 days prior to administration
18. No coagulation abnormality
19. Sign the informed consent statement and voluntarily receive follow-ups, treatments, laboratory tests and other research procedures according to protocol.

Exclusion Criteria:

1. Previous regional or systemic treatment for breast cancer (include but not limited to chemotherapy, radiotherapy, targeted therapy, other clinical trials)
2. Inflammatory breast cancer, bilateral breast cancer or breast cancer already with distant metastasis
3. Complicated with uncontrolled lung disease, severe infection, active peptic ulcer, blood clotting disorders, severe uncontrolled diabetes, connective tissue disorders or bone marrow suppression, and intolerance to neoadjuvant therapy or related treatment
4. Peripheral neuropathy >1 degree caused by any reason
5. History of congestive heart failure, uncontrolled or symptomatic angina, arrhythmias or history of myocardial infarction, refractory hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 100 mmHg);
6. Breast cancer during lactation or pregnancy
7. Unwillingly to receive baseline puncture or neoadjuvant therapy
8. Mental illness or incompliance to treatment caused by other reasons
9. Known history of severe hypersusceptibility to any agents used in the treatment protocol
10. Patients received major surgery or suffered from severe trauma within 2 months of first administration
11. Currently enroll or recently used (30 days within enrollment) other agent under research or involved in other trial
12. Known to be infected with human immunodeficiency virus (HIV)
13. Other circumstances considered to be inappropriate to be enrolled by researchers

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
pathologic Complete Response (pCR) | 3 years
  pCR is defined as the absence of noninvasive tumor residuals in breast and axillary lymph nodes (ypT0/is ypN0) after neoadjuvant therapy.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 3 years
  ORR is defined as the proportion of patients who achieved a complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, MD.PhD., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China